CLINICAL TRIAL: NCT07196540
Title: A Prospective, Non-Randomized, Two-Cohort Clinical Study of Intraperitoneal Injection of Recombinant Modified Human Tumor Necrosis Factor Combined With Tislelizumab and Palliative Radiotherapy in the Treatment of Malignant Ascites From Digestive Tract Tumors After Failure of Previous Standard Treatments
Brief Title: IP rmhTNF-NC + Tislelizumab + Palliat RT for GIT Tumor Malignant Ascites After Failed Std Tx
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, WeiWei Xiao, Chief Physician, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2024-595-01
Record Dates: First submitted 2025-09-15; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Digestive System Neoplasms
MeSH Terms: conditions — Digestive System Neoplasms | interventions — Radiotherapy; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (patients with large-volume abdominal metastatic lesions) (Experimental): Radiotherapy for large-volume abdominal lesions + whole peritoneal cavity low-dose radiotherapy + intraperitoneal infusion (rmhTNF-NC + tislelizumab) Radiotherapy for large-volume abdominal lesions（5-8Gy×5F, D1-D5） whole peritoneal cavity low-dose radiotherapy （1.5Gy×5F, D1-D5） rmhTNF-NC（300IU，ip，D1、D4、 D7、D10） tislelizumab（100mg，ip，D1、D15）
  Interventions: Combination Product: Radiotherapy for large-volume abdominal lesions + whole peritoneal cavity low-dose radiotherapy + rmhTNF-NC + tislelizumab
- Cohort B (patients without measurable abdominal metastatic lesions) (Experimental): Whole peritoneal cavity low-dose radiotherapy + intraperitoneal infusion (rmhTNF-NC + tislelizumab) whole peritoneal cavity low-dose radiotherapy （1.5Gy×5F, D1-D5） rmhTNF-NC（300IU，ip，D1、D4、 D7、D10） tislelizumab（100mg，ip，D1、D15）
  Interventions: Combination Product: Radiotherapy for large-volume abdominal lesions + whole peritoneal cavity low-dose radiotherapy + rmhTNF-NC + tislelizumab

INTERVENTIONS:
Combination Product: Radiotherapy for large-volume abdominal lesions + whole peritoneal cavity low-dose radiotherapy + rmhTNF-NC + tislelizumab — radiotherapy + rmhTNF-NC + tislelizumab

SUMMARY:
This study is a prospective, non-randomized, dual-cohort Phase II clinical trial designed to explore the efficacy and safety of radiotherapy combined with intraperitoneal injection of Recombinant Mutant Human Tumor Necrosis Factor (rmhTNF-NC) and tislelizumab in the treatment of malignant ascites that has failed prior standard therapy.

After completing the informed consent process, eligible patients who meet the inclusion criteria will be enrolled. Participants will receive palliative radiotherapy combined with intraperitoneal perfusion of rmhTNF-NC and tislelizumab according to the study protocol. Before and after one cycle of treatment, abdominal ultrasound will be used to evaluate the response rate of ascites. Safety assessments will be conducted using NCI-CTCAE v5.0.

DETAILED DESCRIPTION:
This study is a prospective, dual-cohort clinical trial following a Simon two-stage design. Eligible subjects who met the inclusion criteria were enrolled. All participants were assigned to the following cohorts, consisting of patients with malignant ascites of the gastrointestinal tract confirmed by cytology or histology, who had experienced failure of prior standard therapy and required clinical intervention due to symptomatic disease. After providing signed informed consent and completing screening procedures, the patients received the following treatments:

Cohort A (patients with large-volume abdominal metastatic lesions):

Radiotherapy for large-volume abdominal lesions + whole peritoneal cavity low-dose radiotherapy + intraperitoneal infusion (rmhTNF-NC + tislelizumab)

Cohort B (patients without measurable abdominal metastatic lesions):

Whole peritoneal cavity low-dose radiotherapy + intraperitoneal infusion (rmhTNF-NC + tislelizumab) All patients received only one treatment cycle. Objective efficacy was evaluated 4 weeks after treatment completion according to WHO criteria. Safety was assessed using NCI-CTCAE version 5.0. Subsequent treatments were not restricted by the study protocol, and clinicians could adjust the treatment plan based on the patient's specific condition.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years, regardless of gender. 2. Histologically or cytologically confirmed malignant ascites originating from digestive system tumors (confirmed by ascites cytology as malignant or clinically diagnosed as peritoneal metastases based on imaging and symptoms).

  3. Presence of large-volume peritoneal metastatic lesions with radiotherapy indications as assessed by a Multidisciplinary Team (MDT) (Cohort A), including an abdominal mass with the longest diameter ≥ 5 cm, or masses invading structures such as the abdominal wall or intra-abdominal muscles causing symptoms like pain.

  4. Moderate or greater amount of ascites, either (first-time treatment) or refractory to previous intraperitoneal therapy with conventional chemotherapeutic agents and/or biological response modifiers. Moderate ascites is defined as: ① Ascites depth ≥ 3 cm on supine ultrasound; ② Accompanied by clinical symptoms (such as chest tightness, shortness of breath, abdominal distension, and discomfort judged by the investigator to be related to ascites).

  5. ECOG performance status of 0-2. 6. Expected survival time > 3 months. 7. Essentially normal cardiac and pulmonary function. 8. Adequate organ function, as evidenced by the following laboratory parameters:
  1. Peripheral blood count: WBC ≥ 4.0 × 10⁹/L, PLT ≥ 80 × 10⁹/L, Hb ≥ 90 g/L.
  2. Renal function: Serum creatinine ≤ 2 × ULN and creatinine clearance (calculated using the Cockcroft-Gault formula) ≥ 40 ml/min.
  3. Liver function: Total bilirubin ≤ 1.5 × Upper Limit of Normal (ULN); or Total bilirubin > ULN but with direct bilirubin ≤ ULN; Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤ 2.5 × ULN (ALT or AST ≤ 5 × ULN allowed for patients with liver metastases).
  4. Adequate coagulation function, defined as an International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 × ULN.

     9. Thyroid Stimulating Hormone (TSH) ≤ ULN; if abnormal, T3 and T4 levels and clinical manifestations should be evaluated; patients can be enrolled if comprehensively assessed and not in an acute active phase.

     10. For non-surgically sterilized or premenopausal female patients, use of a medically approved contraceptive method (e.g., intrauterine device, contraceptive pills, or condoms) is required during the study treatment period and for 6 months after the end of study treatment; Non-surgically sterilized premenopausal female patients must have a negative serum or urine HCG test within 7 days prior to study enrollment; must be non-lactating; For male patients with partners of childbearing potential, effective contraception should be used during the trial and for 6 months after the last dose of the study drug.

     11. Voluntary participation in this study with good compliance, provision of written informed consent, and ability to cooperate with follow-up observations.

     Exclusion Criteria:
* 1. History of allergy to original tumor necrosis factor (TNF), its derivatives, or tislelizumab.

  2. Diagnosis of malignancies other than digestive tract tumor within 5 years prior to the first dose (excluding radically cured basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or carcinoma in situ that has undergone radical resection).

  3. Previous use of tumor necrosis factor (TNF) or its derivative drugs. 4. Significant tumor burden in other organs, and the investigator believes that enrollment in this study would be detrimental to the patient's disease control.

  5. Treatment with any other investigational drugs within 7 days prior to the first dose, or participation in another interventional clinical trial; or receipt of anti-tumor drug therapy (including Chinese herbal medicine with anti-tumor indications) within 7 days before the first dose of the study drug.

  6. Pregnant or breastfeeding women; women of childbearing potential unwilling to use contraception during the study period; or men unwilling to use effective contraception during treatment and for 1 year thereafter.

  7. Significant impairment of vital organ function. 8. Patients with obvious bleeding tendency. 9. Clinically significant or uncontrolled cardiac disease, including unstable angina, acute myocardial infarction within 6 months prior to the first dose, New York Heart Association (NYHA) Class III/IV congestive heart failure, and uncontrolled arrhythmias (subjects with a pacemaker or atrial fibrillation with well-controlled heart rate are allowed).

  10. Presence of ECG changes or history considered clinically significant by the investigator; QTcF interval > 480 ms during screening. For subjects with intraventricular conduction block (QRS interval > 120 ms), JTc interval may be used instead of QTc interval (if JTc is used instead of QTc, JTc must be ≤ 340 ms).

  11. Uncontrolled hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg after optimal medical therapy), history of hypertensive crisis or hypertensive encephalopathy.

  12. Presence of severe acute infection that is uncontrolled; current fever (> 38°C), or presence of purulent and chronic infections, or non-healing wounds.

  13. Patients with radiologically confirmed encapsulated ascites; diagnosed abdominal infection.

  14. Acute or chronic active hepatitis B or C infection: Hepatitis B virus (HBV) DNA > 2000 IU/mL or 10⁴ copies/mL; Hepatitis C virus (HCV) RNA > 10³ copies/mL; co-infection with Hepatitis B surface antigen (HBsAg) and anti-HCV antibody positivity. Subjects can be enrolled if levels are below these criteria after nucleotide antiviral therapy; known history of human immunodeficiency virus (HIV) infection or positive HIV test.

  15. History or evidence of significant bleeding tendency within 3 months prior to enrollment (bleeding > 30 mL, hematemesis, melena, hematochezia within 3 months), hemoptysis (> 5 mL of fresh blood within 4 weeks); history of hereditary or acquired bleeding disorders or coagulation dysfunction; history of clinically significant bleeding symptoms or definite bleeding tendency within 3 months, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, etc.; history of arterial or venous thrombotic diseases within 6 weeks prior to enrollment.

  16. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.

  17. Major surgical procedure (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose of study treatment, or anticipation of the need for major surgery during the study treatment period.

  18. Inadequate recovery from toxicity and/or complications from previous interventions or major surgery prior to initiation of treatment.

  19. Pregnant or lactating women, or subjects who plan to conceive or father children during the study period from screening until the completion of the safety follow-up visit (90 days after the last dose for male subjects).

  20. Radiotherapy within 4 weeks prior to the first dose of the study drug. All radiation-related toxicities must have been resolved, must not require corticosteroids, and must exclude radiation pneumonitis, radiation enteritis, etc. A 2-week washout period is permitted for palliative radiotherapy for non-CNS diseases.

  21. Uncontrolled neurological or psychiatric disorders, or mental disabilities that lead to poor compliance and inability to cooperate or describe treatment response; uncontrolled primary brain tumors or central nervous system metastases with significant symptoms of intracranial hypertension or neuropsychiatric symptoms.

  22. Any other condition deemed by the investigator as inappropriate for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-09-26 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to 4 weeks
  Objective Response Rate (ORR) for Ascites (defined as the proportion of subjects achieving Complete Response (CR) or Partial Response (PR) according to WHO criteria).

IPD SHARING:
Plan to Share IPD: No